CLINICAL TRIAL: NCT03634865
Title: Volar Plates for Distal Radius : Can Epiphyseal Screw Length be Predicted
Brief Title: Screw Lengths in Radius Volar Plates
Acronym: PESLDRF
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PESLDRF (29BRC18.0004)
Record Dates: First submitted 2018-03-08; First posted 2018-08-17 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-02

CONDITIONS: Radius; Fracture, Lower or Distal End; Tendon Injury - Upper Limb; Fracture Fixation, Internal
Keywords: Bone trauma-fracture; Radius; CT-scan; Internal fixation
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background Fractures of the distal radius are among the most common. Major complications, including irritation and rupture of the extensor tendons, may occur if epiphyseal screws of inappropriate length are used.

Questions/Purposes The main objective of the present study was to determine whether the optimal epiphyseal screw length can be determined by reference to the diaphyseal screw length.

Methods Forty CT scans were semi-automatically segmented. A 3D model of the volar plate was affixed to each distal radius with simulation. The maximum lengths of the diaphyseal screws, as well as the four distal epiphyseal screws, were measured. Linear regression analysis was performed.

ELIGIBILITY:
Inclusion Criteria:

* All CT-scans available in our database

Exclusion Criteria:

* Any pathology that could affect the radius morphology
* Refuse to participate

Ages: 17 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that underwent for a CT-Scan of the distal radius from October 2016 to February 2018
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2018-06-06 (Actual); Study Completion 2018-06-06 (Actual)

PRIMARY OUTCOMES:
Main objective | The measures were performed after the CT-Scans were realized. The CT-Scans were performed from October 2016 to February 2018. The measures on the CT-Scans were realized in june 2018
  The main objective of this study was twofold: 1) to assess the anatomical correlation between diaphysis thickness in the diaphyseal screw region of volar plates and epiphyseal thickness in lateral plane with linear regression analysis for each epiphyseal screw length with regard to the diaphysis screw length, and 2) to evaluate whether the optimal epiphyseal screw lengths can be predicted by reference to the diaphyseal screw length when diaphyseal screws are first positioned.
  From the CT-scans, Reconstructions in 3D of the radius were realized. Those reconstructions were used in a computer-simulation study. A Volar plate was affixed to the radius using a specific software.
  Maximum length for each screw located either in epiphysis or diaphysis was measured in mm. This length corresponded with the distance between the entry point of the screw and the opposite point belonging to the wrist along the line perpendicular to the plate.

CONTACTS AND LOCATIONS:
Locations (1):
- CHUR de Brest, Brest, France